CLINICAL TRIAL: NCT02018198
Title: DIStinguish Respiratory Underlying Pathogen associaTed Host Response in Acute Respiratory Infection: An Evaluation of FebriDx POC Test
Brief Title: FebriDx DISRUPT Acute Respiratory Infection Trial in Acute Respiratory Infection: An Evaluation of FebriDx® POC Test
Status: Completed | Type: Observational
Sponsor: Rapid Pathogen Screening (Industry)
Responsible Party: Sponsor
Organization: Lumos Diagnostics (Industry)
Other Study IDs: 13-0830
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Acute Respiratory Tract Infections
Keywords: Host Immune Response; Biomarker; Point-of-Care; Myxovirus Resistance Protein A (MxA); C-reactive Protein (CRP)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Respiratory and blood specimens will be retained for future testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Acute Respiratory Infection: Study subjects will be 1 year of age and older presenting to emergency departments, urgent care centers and primary care offices with a new onset, measured fever and new onset respiratory symptoms.
  Interventions: Diagnostic Test: FebriDx
- Asymptomatic Cohort: Study subjects will be 1 year of age and older presenting to emergency departments, urgent care centers and primary care offices without infection.
  Interventions: Diagnostic Test: FebriDx

INTERVENTIONS:
Diagnostic Test: FebriDx — Point of Care Host Immune Response Test

SUMMARY:
The aim of this study is to determine performance characteristics of the FebriDx test in predicting viral or bacterial infection etiology among febrile (observed or reported) patients presenting the emergency department, urgent care centers or primary care offices with suspected acute respiratory tract infection.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, blinded clinical trial whereby consented study subjects will be enrolled into two study cohorts: an Acute Respiratory Infection cohort and an Asymptomatic cohort. Subjects (children/adolescents, adults and elderly) with suspected community acquired Acute Respiratory Infection will be enrolled in the Acute Respiratory Infection cohort and subjects without infectious illness will be enrolled in the Asymptomatic cohort. All subjects will undergo FebriDx testing (study device) and results, blinded to subjects and treating physicians, will be compared to a Clinical Reference Algorithm supervised by clinical experts to arbitrate the presence and type of infection (bacterial or viral); the experts are also blinded to the results of FebriDx testing.

The FebriDx® test is a rapid, point-of-care (POC) test that uses a fingerstick blood sample to identify patients with a pathogen induced host immune response through in-vitro detection of both Myxovirus resistance protein A (MxA) and c-reactive protein (CRP) directly from a whole blood sample. MxA is an intracellular protein that becomes elevated in the presence of acute viral infection and CRP is an acute-phase inflammatory protein that is elevated in the presence of a systemic bacterial and/or viral infection.

ELIGIBILITY:
Acute Respiratory Infection Cohort INCLUSION CRITERIA

* 1 year of age or older
* Exhibit or report of a new onset measured temperature (oral or tympanic) of greater than or equal to 100.5°F/38°C within 3 days (72 hours) of enrollment
* Clinical suspicion for Acute Respiratory Infection and presents with at least one of the following new onset of symptoms: runny nose, nasal congestion, sore throat, cough, hoarse voice or shortness of breath beginning within 7 days before enrollment

Acute Respiratory Infection Cohort EXCLUSION CRITERIA

* Incomplete or invalid testing for comparator method
* Unwilling to participate
* Receiving interferon therapy (e.g. MS, HIV, HBV, HCV) in the last 30 days
* Immunocompromised state (e.g. HIV) or taking immunosuppressive or chemotherapeutic medications in the last 30 days (e.g. oral steroids, Methotrexate, Cyclosporine, Antimetabolite chemotherapy, interferon therapy)
* Taking antibiotics or antiviral therapy in the last 14 days
* Received a live viral immunization in the last 14 days
* Significant trauma or burns (> 5% total body surface area or full thickness (3rd°)) in the last 30 days
* Major surgery (requiring intravenous anesthesia and/or respiratory assistance) in the last 30 days
* Chronic fever without associated respiratory symptoms of greater than 7 days
* History of ear pain plus an exam consistent with otitis media within the last 14 days
* History of a myocardial infarction or stroke in the last 30 days

ASYMPTOMATIC COHORT INCLUSION CRITERIA

* 1 year of age or older
* Absence of infectious signs and symptoms

ASYMPTOMATIC COHORT EXCLUSION CRITERIA

* Fever greater than or equal to 100.5°F /38°C (oral or tympanic) in last 14 days
* Cough
* Chills
* Dyspnea
* Purulent Sputum
* Fatigue
* Pleuritic Pain
* Nasal congestion
* Rhinorrhea (runny nose)
* Sore throat
* Hoarse voice
* Earache
* Autoimmune or rheumatologic disease (e.g. undifferentiated connective tissue disease, Rheumatoid Arthritis, Systemic Lupus Erythematosus (and subsets of Lupus), Sjögren's syndrome, Systemic Sclerosis, Polymyositis and Dermatomyositis, Wegener's granulomatosis)
* Suspected of having any infection
* Receiving interferon therapy (e.g. MS, HIV, HBV, HCV) in last 30 days
* Immunocompromised state (e.g. HIV) or taking immunosuppressive (e.g. oral steroids, Methotrexate, Cyclosporine, Antimetabolite chemotherapy, interferon therapy) in the last 30 days
* Taking antibiotics or antiviral therapy in the last 30 days
* Received a live viral immunization in the last 30 days
* Significant trauma or burns (> 5% total body surface area or full thickness (3rd°)) in the last 30 days
* Major surgery (requiring intravenous anesthesia and/or respiratory assistance) in the last 30 days
* History of a myocardial infarction or stroke in the last 30 days
* Chronic bacterial infection or osteomyelitis
* Known chronic viral infections such as HIV, HCV, HBV, or CMV
* Active tuberculosis
* Acute or chronic (greater than 30 days) diarrhea and/or vomiting
* Urinary tract symptoms in the last 14 days
* Active diarrheal illness within the last 14 days
* Active skin, ocular, or neurologic infections
* Suspected of having otitis media

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with a new onset, measured fever (exhibited or reported) and acute respiratory symptoms
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the presence of a bacterial associated systemic host immune response or viral associated systemic host immune response related to an acute community acquired febrile acute respiratory tract infection, as compared to final diagnosis | 10 minutes
  The primary analysis will determine performance characteristics of the FebriDx® test by assessing negative and positive agreement of the FebriDx® results in determining the presence of a bacterial associated systemic host immune response or viral associated systemic host immune response compared with a Clinical Reference Algorithm (comparator method) that is supervised by clinical experts.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Shapiro, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (20):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - AFC Urgent Care/Urgent Care Clinical Trials, Denver, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Doral Medical Research, Hialeah, Florida
  - PAS Research, Tampa, Florida
  - Massachusetts General, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Vincent Hospital, Worcester, Massachusetts
  - New York Methodist Hospital, Brooklyn, New York
  - Woodruff Road Urgent Care Center/Urgent Care Clinical Trials, Easley, South Carolina
  - Parkside Pediatrics, Greenville, South Carolina
  - Woodruff Road Urgent Care Center, P.C./ Urgent Care Clinical Trials, Greenville, South Carolina
  - AFC Urgent Care/Urgent Care Clinical Trials, Chattanooga, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - VA Office of Research and Development/Vanderbilt University School of Medicine, Nashville, Tennessee
  - Urgent Care Clinical Trials, Dallas, Texas
  - Benchmark Research, San Angelo, Texas
  - University of Wisconsin-Madison/Berbee Walsh Department of Emergency Medicine, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joseph P, Godofsky E. Outpatient Antibiotic Stewardship: A Growing Frontier-Combining Myxovirus Resistance Protein A With Other Biomarkers to Improve Antibiotic Use. Open Forum Infect Dis. 2018 Feb 15;5(2):ofy024. doi: 10.1093/ofid/ofy024. eCollection 2018 Feb. PMID 29479553
- [Result] Shapiro NI, Self WH, Rosen J, Sharp SC, Filbin MR, Hou PC, Parekh AD, Kurz MC, Sambursky R. A prospective, multi-centre US clinical trial to determine accuracy of FebriDx point-of-care testing for acute upper respiratory infections with and without a confirmed fever. Ann Med. 2018 Aug;50(5):420-429. doi: 10.1080/07853890.2018.1474002. Epub 2018 May 18. PMID 29775092
- [Result] Self WH, Rosen J, Sharp SC, Filbin MR, Hou PC, Parekh AD, Kurz MC, Shapiro NI. Diagnostic Accuracy of FebriDx: A Rapid Test to Detect Immune Responses to Viral and Bacterial Upper Respiratory Infections. J Clin Med. 2017 Oct 7;6(10):94. doi: 10.3390/jcm6100094. PMID 28991170
- [Result] Shapiro NI, Filbin MR, Hou PC, Kurz MC, Han JH, Aufderheide TP, Ward MA, Pulia MS, Birkhahn RH, Diaz JL, Hughes TL, Harsch MR, Bell A, Suarez-Cuervo C, Sambursky R. Diagnostic Accuracy of a Bacterial and Viral Biomarker Point-of-Care Test in the Outpatient Setting. JAMA Netw Open. 2022 Oct 3;5(10):e2234588. doi: 10.1001/jamanetworkopen.2022.34588. PMID 36255727